CLINICAL TRIAL: NCT05447286
Title: Clinical Evaluation of NMDA Modulator NYX-783 for OUD: Randomized, Double-blind, Placebo-Controlled Study to Assess Safety, Tolerability, and Pharmacokinetics of NYX-783 in Combination With Oxycodone (Study 1)
Brief Title: Safety, Tolerability and Pharmacokinetics of NYX-783 and Oxycodone DDI Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, RAJITA SINHA, PROFESSOR, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000033008; UG3DA050322 (NIH); NYX-783-1009 (Other: Aptinyx)
Record Dates: First submitted 2022-06-21; First posted 2022-07-07 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo + Oxycodone (Placebo Comparator): Participants will receive placebo with + 15 mg oxycodone then placebo + 30 mg oxycodone in separate inpatient randomized sessions in this, cross-over study over 6 experimental sessions.
  Interventions: Drug: Placebo; Drug: Oxycodone
- NYX-783: 50 mg dose + Oxycodone (Active Comparator): Participants will receive NYX-783 50 mg dose with + 15 mg oxycodone then NYX-783 50 mg + 30 mg oxycodone in separate inpatient randomized sessions in this, cross-over study over 6 experimental sessions.
  Interventions: Drug: NYX-783; Drug: Oxycodone
- NYX-783: 150 mg dose + Oxycodone (Active Comparator): Participants will receive NYX-783 150 mg dose with + 15 mg oxycodone then NYX-783 150 mg + 30 mg oxycodone in separate inpatient randomized sessions in this, cross-over study over 6 experimental sessions.
  Interventions: Drug: NYX-783; Drug: Oxycodone

INTERVENTIONS:
Drug: NYX-783 — This study proposes to examine the safety, tolerability, and pharmacokinetics (PK) of NYX-783 at 50 mg and 150 mg doses versus Placebo (PBO) in combination with acute Oxycodone 15 mg and 30 mg in an inpatient randomized, cross-over study over 6 experimental sessions.
  Other Names: ((2S, 3R)-3-hydroxy-2-((S)-5-isobutyryl-1-oxo-2,5-diazaspiro[3.4]octan-2-yl)butanamide)
  Arms: NYX-783: 150 mg dose + Oxycodone; NYX-783: 50 mg dose + Oxycodone
Drug: Placebo — This study proposes to examine the safety, tolerability, and pharmacokinetics (PK) of NYX-783 at 50 mg and 150 mg doses versus Placebo (PBO) in combination with acute Oxycodone 15 mg and 30 mg in an inpatient randomized, cross-over study over 6 experimental sessions.
  Arms: Placebo + Oxycodone
Drug: Oxycodone — This study proposes to examine the safety, tolerability, and pharmacokinetics (PK) of NYX-783 at 50 mg and 150 mg doses versus Placebo (PBO) in combination with acute Oxycodone 15 mg and 30 mg in an inpatient randomized, cross-over study over 6 experimental sessions.

SUMMARY:
This study proposes to examine the safety, tolerability, and pharmacokinetics (PK) of NYX-783 50 mg and 150 mg versus Placebo (PBO) in combination with acute Oxycodone 15 mg and 30 mg in an inpatient randomized, cross-over study in non-treatment seeking non-dependent, opioid experienced individuals with current recreational use.

DETAILED DESCRIPTION:
Outcomes will be cardiovascular (ECG monitoring, heart rate, blood pressure), respiratory, Clinical Opioid Withdrawal Scale (COWS), treatment emergent adverse events (TEAEs), and PK of NYX-783 levels in combination with Oxycodone. Secondary outcomes will be drug effects, subjective opiate withdrawal scale (SOWS), Drug Effects Questionnaire (DEQ), pupillary diameter, the Opioid Symptom Checklist (OSC), craving, stress and pain, and study drug levels during NYX-783 and Oxycodone combination challenge sessions.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, written, informed consent.
* full scale and verbal IQs > 80 (Shipley Institute of Living IQ Screening Test).
* Non-treatment seeking, non-dependent, opioid-experienced participants with low, opioid use via smoking or oral pills routes and with no need for medical detoxification from opiates and without past 12-month history of overdoses or medical detoxification for opioid withdrawal.
* Participants must agree to use dual contraceptive methods during the study and refrain from donating sperm or ova during study or for 28 days after final dose of drug for ova and for 90 days after final dose of drug for sperm. Dual contraceptive methods include the use of a barrier contraceptive (i.e., condoms) in addition to another effective method that can prevent pregnancy (i.e., oral or parenteral contraceptives, intrauterine devices, spermicide, etc.).
* Ability to understand and comply with study requirements and restrictions and provide a secondary contact if they cannot be reached.

Exclusion Criteria:

* Meet current DSM-5 criteria of moderate to severe Substance Use Disorder (SUD) on either sedative, hypnotics, cocaine, methamphetamine, opiates or alcohol.
* Daily heroin, fentanyl use requiring opiate detoxification and treatment.
* Regular daily prescribed use of anticonvulsants, sedatives/hypnotics, other antihypertensives, anti-arrhythmics, antiretroviral medications, naltrexone, antabuse, grapefruit juice and St. John's wort products, glucocorticoids, stimulants (amphetamine like compounds), CNS active medications (other than stabilized use of antidepressants and anti-anxiety medications), metformin, or other medications such as benzodiazepines and sedating antidepressants that in the opinion of the investigators interfere with the study.
* Women who are pregnant or nursing (as assessed by pregnancy tests during initial intake and upon CNRU admissions).
* HIV seropositivity, hepatitis or other acute ongoing infectious disease considered clinically significant by the investigator.
* Traumatic brain injury with loss of consciousness.
* Individuals with current or past history of seizure disorders.
* Current or recent diagnosis within past 6-months of Major Depressive Disorder (MDD), bipolar disorder, schizophrenia, and schizoaffective disorder.
* History of a neurodegenerative or neuro-inflammatory disorder including Huntington's, Parkinson's, Alzheimer's disease, or multiple sclerosis.
* Known familial history or known presence of long QT syndrome, or a known history of past or current clinically significant arrhythmias or ischemic heart disease.
* History of gastrointestinal disease or surgery (except simply appendectomy or hernia repair), leading to impaired drug absorption.
* Uncorrected hypothyroidism or hyperthyroidism. Participants with compensated hypothyroidism with normal thyroid-stimulating hormone levels may be enrolled.
* Sensitivity, allergy, or intolerance to N-methyl-D-aspartate receptor (NMDAR) ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone and magnesium. Use of NMDAR-binding drugs within 60 days prior to dosing or during the study.
* Received an investigational product or device within 30 days of dosing (or 5 half-lives whichever is longer).
* Previously received NYX-783.
* Screening QT interval corrected for heart rate (HR) by Fridericia's formula (QTcF) > 450 (males) or 470 (females) milliseconds (msec) or an ECG that is not suitable for QT measurements (e.g., poorly defined termination of T-wave in the investigator's opinion.
* Heart rate ≤45 or >90 bpm at screening
* Creatinine clearance <60ml/min at screening or history of renal disease as assessed by Investigator.
* Uncontrolled Type I or Type II diabetes or uncontrolled hypertension characterized by fasting blood glucose > 126 mg/dl or postprandial blood glucose > 200 mg/dl, resting systolic blood pressure >160 mm Hg or resting diastolic >100 mm Hg, or clinically significant hypotension in the judgement of the Investigator as characterized by resting systolic blood pressure <90 mm Hg or resting diastolic blood pressure <60 mm Hg.
* Impaired hepatic function characterized by a previous known diagnosis of chronic liver disease and/or the presence of:

  1. direct bilirubin > 1.5x the upper limit of normal at screening
  2. alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase, or gamma-glutamyl transferase (GGT) > 2x the upper limit of normal at screening.
* History of severe COVID-19 infection requiring hospitalization, treatment with oxygen or mechanical ventilation, that may interfere with study participation as assessment by the Investigator.
* Any participant with a medical history of Covid-19 infection (positive test) within the last 2 months, or current symptoms consistent with Covid-19 infection, as assessed by the Investigator.
* Donated blood during the past 8 weeks.
* Participants who do not report an increase in subjective opioid effect, as measured by the Drug Effects Questionnaire (DEQ, see below) by minimum of 10% or more to initial challenge with oxycodone in Session 1 will be excluded from the DDI phase sessions 2-7.

Ages: 21 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in respiratory rate | over 6 sessions from baseline up to 3 weeks
  Change in respiratory rate pre and post drug administration measured by counting breaths
Change in oxygenation saturation | over 6 sessions from baseline up to 3 weeks
  Change in oxygenation saturation pre and post drug administration measured by pulse-oximeter
Change in blood pressure | over 6 sessions from baseline up to 3 weeks
  Change in blood pressure pre and post drug administration measured by blood pressure monitor
Change in heart rate | over 6 sessions from baseline up to 3 weeks
  Change in heart rate pre and post drug administration measured by blood pressure monitor
Change in body temperature | over 6 sessions from baseline up to 3 weeks
  Change in body temperature pre and post drug administration measured by temperature monitor
Change in cardiac rate | over 6 sessions from baseline up to 3 weeks
  Change in cardiac rate pre and post drug administration measured by EKG cardiac monitor
Change in cardiac rhythm | over 6 sessions from baseline up to 3 weeks
  Change in cardiac rhythm pre and post drug administration measured by EKG cardiac monitor

SECONDARY OUTCOMES:
treatment emergent adverse events (TEAES) from Systematic Assessment for Treatment Emergent Effects (SAFTEE) | over 6 sessions from baseline up to 3 weeks
  The SAFTEE is a technique for the systematic assessment of side effects in clinical trials that rates the current severity of a wide range of somatic, behavioral and affective symptoms and tabulates occurrence of each TEAE symptom
Change in Clinical Opiate Withdrawal Scale (COWS) | over 6 sessions from baseline up to 3 weeks
  COWS is an 11-item scale to rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. The summed score determines the stage/severity of opiate withdrawal and assess the level of physical dependence on opioids. Score: 5- 12 = mild; 13-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal
Change in Subjective Opioid Withdrawal Scale (SOWS) | over 6 sessions from baseline up to 3 weeks
  SOWS is a self-administered scale for opioid withdrawal symptoms. It has16 symptoms whose intensity is rated on a scale of 0 (not at all) to 4 (extremely). Mild Withdrawal = score of 1-10, Moderate withdrawal = 11-20, Severe withdrawal = 21-30
Change in Drug Effects Questionnaire (DEQ) | over 6 sessions from baseline up to 3 weeks
  The DEQ measures Good Drug Effect and consists of 11 questions with total score range from 0-100. Higher scores indicate more positive effects.
Change in Visual Analog Scale (VAS) | over 6 sessions from baseline up to 3 weeks
  The VAS scales are 5 item drug effect self report ratings The visual analog questions were "Do you feel any Drug Effect?" "Do you like the drug?" "How high are you?" "Does the drug have any Good Effects?" "Does the drug have any Bad Effects?" and "How much do you DESIRE opiates?" The subjects responded by positioning an arrow along a 100-point line labeled with "not at all" at one end and "extremely" at the other. High scores show drug effect and craving, low scores show low drug effect and low craving
Change in Opioid Symptom Checklist (OSC) | over 6 sessions from baseline up to 3 weeks
  The OSC is a 13-item opioid symptom checklist consisting of true/false questions designed to measure opioid effects (e.g., "My skin is itchy"). True scores total up to acute opiate positive and negative symptoms and low true scores will mean not feeling any of the negative and positive symptoms.
Change in pupillary diameter | over 6 sessions from baseline up to 3 weeks
  pupil diameter size using pupilometer

OTHER OUTCOMES:
Pharmacokinetic (PK) levels of study medication | across 3 sessions during the 3 weeks assessment period
  plasma levels drawn repeatedly in 3 experimental sessions

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Cmhc/Cnru, New Haven, Connecticut
  - The Yale Stress Center: Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No